CLINICAL TRIAL: NCT06106958
Title: The Effects of Foot Rehabilitation And Minimalist Shoes (FRAMES) on Pain, Strength, and Function in Adults With Plantar Fasciopathy
Brief Title: Effects of Foot Rehabilitation And Minimalist Shoes on Pain, Strength, and Function in Adults With Plantar Fasciopathy
Acronym: FRAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jen Xu, Doctoral Student, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSR230045
Record Dates: First submitted 2023-10-19; First posted 2023-10-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Plantar Fascitis; Plantar Fasciopathy; Plantar Fasciitis of Both Feet; Plantar Fasciitis of Right Foot; Plantar Fasciitis of Left Foot; Plantar Fasciitis, Chronic
Keywords: plantar fasciitis; intrinsic foot muscles; minimalist shoes
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: There will be two groups:
  1. Performing foot rehabilitation exercises and wearing minimalist shoes (intervention group)
  2. Only performing foot rehabilitation exercises (control group)
Who Masked: Outcomes Assessor
Masking Description: The investigator assessing laboratory-based outcome measures will be blinded to group allocation and will not be the member of the study team communicating with participants about their intervention protocols.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foot Rehabilitation And Minimalist Shoes (FRAMES) (Experimental): The intervention group will receive a pair of minimalist shoes along with a home exercise program and a protocol that indicates how to slowly adjust to wearing the shoes.
  Interventions: Behavioral: Home Exercise Program; Behavioral: Minimalist Shoes
- Home Exercise Program (Control) (Active Comparator): The intervention group will receive a home exercise program.
  Interventions: Behavioral: Home Exercise Program

INTERVENTIONS:
Behavioral: Home Exercise Program — Participants will receive a home exercise program that consists of 2 exercises and 3 stretches. The exercises include:
  * Massage on the bottom of the foot with a ball
  * Calf-raises
  * Lunge calf-stretch with the knee straight
  * Calf-stretch with the knee bent
  * Stretch for the bottom of the foot
  These exercises are intended to be performed daily.
Behavioral: Minimalist Shoes — Participants will receive a pair of minimalist shoes. They will wear them for an allotted amount of time per day each week, in order to allow for a slow adjustment into the shoes. The protocol is as follows:
  * Week 1: 1 hour per day
  * Week 2: 2 hours per day
  * Week 3: 4 hours per day
  * Week 4: 6 hours per day
  * Week 5: 8 hours per day
  * Week 6: 8 hours per day
  * Week 7: 8 hours per day
  * Week 8: 8 hours per day
  Arms: Foot Rehabilitation And Minimalist Shoes (FRAMES)

SUMMARY:
The goal of this clinical trial is to compare the effects of 8 weeks of foot rehabilitation exercises in conjunction with wearing minimalist shoes in individuals with plantar fasciopathy, compared to only performing foot rehabilitation exercises. The main questions it aims to answer are:

* Will individuals with plantar fasciopathy be able to reduce their pain and improve their self-reported function by performing rehabilitation exercises and wearing minimalist shoes, compared to those only performing rehabilitation exercises?
* Will individuals with plantar fasciopathy be able to increase their intrinsic foot muscle strength and size, their balance, and gait biomechanics by performing rehabilitation exercises and wearing minimalist shoes, compared to those only performing rehabilitation exercises?
* What characteristics of individuals with plantar fasciopathy make them most suited to succeed in a protocol of performing rehabilitation exercises and wearing minimalist shoes?

Participants will be asked to come into the lab at the start of the intervention and after 8 weeks, where the following will be assessed:

* Patient-reported outcomes
* Foot morphology
* Intrinsic foot muscle strength
* Balance
* Gait biomechanics

For the intervention, participants in both groups will perform the same rehabilitation exercises, including:

* Massage to the bottom of the foot
* Calf-raises
* Calf and foot stretches

DETAILED DESCRIPTION:
The purpose of the study is to determine the effects of 8-weeks of wearing minimalist shoes and performing a home exercise program (intervention group) on pain, self-reported function, intrinsic foot muscle strength and size, balance, and gait biomechanics, as opposed to receiving a home exercise program alone (control group).

All participants will report to the Exercise and Sport Injury Laboratory for a baseline clinical assessment performed by a blinded assessor to determine their level of pain and their self-reported function using a variety of patient-reported outcomes. These include pain levels on a Visual Analog Scale (VAS), Global Rating of Change to assess perceived changes in function, Foot Health Status Questionnaire (FHSQ) to gather general and foot-related health information, and a variety of scales that assess kinesiophobia, fear-avoidance belief, self-efficacy, and activity level. Functional measures include intrinsic foot muscle strength via diagnostic ultrasound, intrinsic foot muscle size via two different types of handheld dynamometer, balance via a single-leg balancing task on a force plate, and gait biomechanics via a walking task with insoles that can obtain measures of force and loading rate.

At the end of the first baseline visit, all participants will be taught how to perform the home rehabilitation exercise routine, and handed an informational sheet that will have pictures and links to supplemental videos to ensure that they understand the exercises and have the resources to review.

Immediately following the first baseline visit, participants will meet with another member of the study team to ensure assessor blinding. They will be randomly assigned to one of two groups: the intervention group of foot rehabilitation and minimalist shoes (intervention), or the control group of just rehabilitation exercises (control). The randomization sequence will be created a priori with a random-number generator stratified by sex, placed in sealed opaque envelopes by another member of the study team to blind the assessor. Participants in the intervention group will have a pair of shoes ordered for them, and they will begin the protocol when the shoes have arrived.

Participants in both groups will be instructed to fill out a daily survey that will be sent via text and stored in a secure server (REDCap), that will indicate if they have completed their rehabilitation exercises. Participants will also all wear Fitbit smart watches that will track their step count and some other health-related metrics. They will not be able to see their own data during the protocol.

At the 4-week mark of the study, all individuals will be sent a link to take surveys of patient-reported outcomes, including pain levels, self-reported function, kinesiophobia, fear-avoidance belief, self-efficacy, and activity level. They will also complete a phone call with a member of the study team (not the assessor, to maintain blinding) as a check-in to discuss pain levels and any other questions and concerns they have.

At the end of the 8-weeks, individuals will return to the lab to have the same measures as the baseline session completed. The investigators will then be able to determine if performing foot rehabilitation exercises and wearing minimalist shoes reduces pain, improves self-reported function, and increases intrinsic foot muscle strength and size, balance, and gait biomechanics, compared to baseline and to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18 - 55 years old
* First-step pain in the morning over past week - Visual Analog Score between 30-70 mm
* Heel pain for at least a month with an insidious onset

Exclusion Criteria:

* Other current lower extremity neuromusculoskeletal injury
* Other lower extremity neuromusculoskeletal injuries other than the foot in the past 3 months
* Previous history of foot/ankle fractures or surgeries
* Current participation in formal rehab for plantar fasciopathy
* Previous minimalist shoe experience

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Pain | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Visual Analog Scale (0-100 mm) pain outcome scores for the following items:
  * Average pain over the past week
  * First-step pain over the past week (the pain that is felt upon waking up in the morning and taking a first step)
  * Average heel pain of the day
Change in perception of overall recovery | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Global Rating of Change (GROC) outcome scores
Change in self-reported function and health | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Foot Health Status Questionnaire (FHSQ) outcome scores
Change in foot morphology: length, width, arch height, and girth | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Arch Height Index tool outcome measures
Change in intrinsic foot muscle size | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Muscle thickness and cross-sectional area of the abductor hallucis, flexor hallucis brevis, flexor digitorum brevis, and quadratus plantae, using diagnostic ultrasound in a weight-bearing position.
Change in intrinsic foot muscle strength | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Tested separately for the great toe and lesser toes using two different types of handheld dynamometer
Change in center of pressure (COP) distance during balance | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  COP distance using a force plate during a single-limb balance task, eyes open and eyes closed.
Change in foot posture outcomes | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Clinical foot posture index assessment (23-point scale)
Change in center of pressure (COP) velocity during balance | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  COP velocity using a force plate during a single-limb balance task, eyes open and eyes closed.
Change in center of pressure (COP) 95% ellipse area during balance | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  COP 95% ellipse area using a force plate during a single-limb balance task, eyes open and eyes closed.
Change in vertical ground reaction force (vGRF) of the rearfoot | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The force (N) during treadmill and overground walking using loadsol sensors

SECONDARY OUTCOMES:
Change in kinesiophobia | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Tampa Scale of Kinesiophobia (TSK-11) outcome scores
Change in fear-avoidance belief | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Fear-Avoidance Belief Questionnaire (FABQ) outcome scores
Change in pain self-efficacy | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  Pain Self-Efficacy Questionnaire (PSEQ) outcome scores
Change in activity level | This outcome change will be measured from baseline, to the midpoint of the intervention (4 weeks), to the end of the intervention (8 weeks) for both groups.
  National Aeronautics and Space Administration Activity Survey (NAS)
Change in vertical ground reaction force (vGRF) of the whole foot | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The force (N) during treadmill and overground walking using loadsol sensors
Change in vertical ground reaction force (vGRF) of the midfoot | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The force (N) during treadmill and overground walking using loadsol sensors
Change in vertical ground reaction force (vGRF) of the forefoot | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The force (N) during treadmill and overground walking using loadsol sensors
Change in average loading rate | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The loading rate (N/s) during treadmill and overground walking using loadsol sensors
Change in instantaneous loading rate | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  The loading rate (N/s) during treadmill and overground walking using loadsol sensors
Change in knee sagittal plane kinematics | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Knee sagittal plane joint moment (in Nm/kg) measured during the overground gait analysis using markerless motion capture
Change in hip sagittal plane kinematics | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Hip sagittal plane joint moment (in Nm/kg) measured during the overground gait analysis using markerless motion capture
Change in ankle sagittal plane kinematics | This outcome change will be measured from baseline, to the end of the intervention (8 weeks) for both groups.
  Ankle sagittal plane joint moment (in Nm/kg) measured during the overground gait analysis using markerless motion capture
Change in steps per day | This outcome change will be measured everyday for 8 weeks
  Steps per day measured on a Fitbit
Change in activity level per day | This outcome change will be measured everyday for 8 weeks
  Hours of activity per day measured on a Fitbit

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Xu, MS, Principal Investigator — University of Virginia; Susan Saliba, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnes A, Sullivan J, Pappas E, Adams R, Burns J. Clinical and Functional Characteristics of People With Chronic and Recent-Onset Plantar Heel Pain. PM R. 2017 Nov;9(11):1128-1134. doi: 10.1016/j.pmrj.2017.04.009. Epub 2017 Apr 28. PMID 28461226
- [Background] Allen RH, Gross MT. Toe flexors strength and passive extension range of motion of the first metatarsophalangeal joint in individuals with plantar fasciitis. J Orthop Sports Phys Ther. 2003 Aug;33(8):468-78. doi: 10.2519/jospt.2003.33.8.468. PMID 12968860
- [Background] Cheung RT, Sze LK, Mok NW, Ng GY. Intrinsic foot muscle volume in experienced runners with and without chronic plantar fasciitis. J Sci Med Sport. 2016 Sep;19(9):713-5. doi: 10.1016/j.jsams.2015.11.004. Epub 2015 Nov 22. PMID 26655866
- [Background] Chang R, Rodrigues PA, Van Emmerik RE, Hamill J. Multi-segment foot kinematics and ground reaction forces during gait of individuals with plantar fasciitis. J Biomech. 2014 Aug 22;47(11):2571-7. doi: 10.1016/j.jbiomech.2014.06.003. Epub 2014 Jun 11. PMID 24992816
- [Background] Wearing SC, Smeathers JE, Urry SR, Hennig EM, Hills AP. The pathomechanics of plantar fasciitis. Sports Med. 2006;36(7):585-611. doi: 10.2165/00007256-200636070-00004. PMID 16796396
- [Background] Jaffri AH, Koldenhoven R, Saliba S, Hertel J. Evidence for Intrinsic Foot Muscle Training in Improving Foot Function: A Systematic Review and Meta-Analysis. J Athl Train. 2023 Nov 1;58(11-12):941-951. doi: 10.4085/1062-6050-0162.22. PMID 35724360
- [Background] Newsham K. Exploring Workload Associated With Learning Foot Core Exercises. International Journal of Athletic Therapy and Training. 2022;27(3):120-128.
- [Background] Ridge ST, Olsen MT, Bruening DA, Jurgensmeier K, Griffin D, Davis IS, Johnson AW. Walking in Minimalist Shoes Is Effective for Strengthening Foot Muscles. Med Sci Sports Exerc. 2019 Jan;51(1):104-113. doi: 10.1249/MSS.0000000000001751. PMID 30113521
- [Background] Warne JP, Gruber AH. Transitioning to Minimal Footwear: a Systematic Review of Methods and Future Clinical Recommendations. Sports Med Open. 2017 Sep 15;3(1):33. doi: 10.1186/s40798-017-0096-x. PMID 28916956
- [Background] Ribeiro AP, Joao SMA. The Effect of Short and Long-Term Therapeutic Treatment with Insoles and Shoes on Pain, Function, and Plantar Load Parameters of Women with Plantar Fasciitis: A Randomized Controlled Trial. Medicina (Kaunas). 2022 Oct 28;58(11):1546. doi: 10.3390/medicina58111546. PMID 36363506
- [Background] Yeasmin Lipa L, Kalita A, Dutta A. A Comparative Study To Find Out The Effectiveness Of Myofascial Release Technique Along With Stretching Versus Myofascial Release Technique In Patients With Plantar Fasciitis. Int J Life Sci Pharm Res. Published online January 31, 2022. doi:10.22376/ijpbs/lpr.2022.12.1.L183-193
- [Background] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Background] Campitelli NA, Spencer SA, Bernhard K, Heard K, Kidon A. Effect of Vibram FiveFingers Minimalist Shoes on the Abductor Hallucis Muscle. J Am Podiatr Med Assoc. 2016 Sep 2;106(5):344-351. doi: 10.7547/14-084. PMID 27762613
- [Background] Kamonseki DH, Goncalves GA, Yi LC, Junior IL. Effect of stretching with and without muscle strengthening exercises for the foot and hip in patients with plantar fasciitis: A randomized controlled single-blind clinical trial. Man Ther. 2016 Jun;23:76-82. doi: 10.1016/j.math.2015.10.006. Epub 2015 Oct 30. PMID 26654252